CLINICAL TRIAL: NCT02055664
Title: THE TAP BLOCK TECHNIQUE VIA THE ANTERIOR APPROACH IN ELECTIVE SURGERY OF THE SPINE: Prospective, Randomised, Double Blind Trial, Comparing TAP BLOCK With Continuous Infiltration of Ropivacaine Versus Placebo
Brief Title: The Tap Block Technique Via the Anterior Approach in Elective Surgery of the Spine
Acronym: TAPBloc Rachis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: MIREK 2013
Record Dates: First submitted 2014-02-04; First posted 2014-02-05 (Estimated); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Elective Surgery of the Spine by Laparotomy

ARMS (2):
- treatment (Experimental)
  Interventions: Drug: Chlorure de sodium 0.9%
- control (Placebo Comparator)
  Interventions: Drug: Ropivacaine 0.2%

INTERVENTIONS:
Drug: Ropivacaine 0.2%
  Arms: control
Drug: Chlorure de sodium 0.9%
  Arms: treatment

SUMMARY:
This is a prospective, single-centre, randomised, double-blind trial, comparing TAP block with continuous infiltration of ropivacaine versus placebo.

Procedure:

Once consent has been obtained, patients will be randomised into one of the two groups: Ropivacaine or Placebo. At the end of the operation, the TAP block will be implemented via a catheter inserted by the anaesthetist.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 yo who have provided written informed consent
* Patients with an indication for elective spinal surgery using laparotomy
* Patients with national health insurance cover

Exclusion Criteria:

* Adults under guardianship
* Pregnant or breast-feeding women
* allergies or contra-indication for paracetamol, morphine-based drugs
* Contra-indication for ropivacaine
* Contra-indication for sodium chloride
* inability to understand PCA (patient-controlled anaesthesia)
* Hypersensitivity to ropivacaine or to other aminoamide local anaesthetics
* Hypovolemia

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-01-23 (Actual); Primary Completion 2015-08-12 (Actual)

PRIMARY OUTCOMES:
Consumption of morphine in mg | First 48 hours following the surgery

SECONDARY OUTCOMES:
Intensity of pain | First 48 hours following the surgery

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Dijon, Dijon, France